CLINICAL TRIAL: NCT06329063
Title: Vasopressin Modulates Neural Responses to Looming Visual Stimuli: An Eye-tracking Study
Brief Title: Oral Vasopressin Modulates Neural Responses to Looming Visual Stimuli: An Eye-tracking Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BAM_lab_eyetracking_03
Record Dates: First submitted 2024-03-15; First posted 2024-03-25 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Eye-tracking; vasopressin; looming fear
MeSH Terms: conditions — Diabetes Insipidus | interventions — Vasopressins

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomized placebo-controlled double-blind between-subject design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vasopressin group (Experimental): Drug: Vasopressin (20IU)
  Interventions: Drug: Vasopressin
- Placebo group (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vasopressin — Administration of vasopressin (20 IU) (oral spray)
  Other Names: Antidiuretic Hormone
  Arms: Vasopressin group
Drug: Placebo — Administration of placebo (oral spray)
  Other Names: Placebo treatment
  Arms: Placebo group

SUMMARY:
The main aim of the present study is to investigate the effects of orally administered vasopressin (AVP) on the perception of time-to-collision of threatening and non-threatening stimuli by combining a validated looming fear eye-tracking paradigm with a randomized between-subject placebo-controlled pharmacological trial design.

DETAILED DESCRIPTION:
Animal models and initial findings in humans suggest a role of the AVP signaling system in socio-emotional processes. At the same time, the visual system's remarkable ability to perceive and interpret impending threats, notably through the "looming" phenomenon- a distinct pattern of optical expansion on the retina as objects approach, theoretically allows for precise estimation of the time-to-collision (TTC). It was recently demonstrated that the affective content of looming stimuli influences perceived TTC, with threatening objects judged as approaching sooner than non-threatening objects, hinting at a nuanced interaction between emotional valence and temporal perception. Within this context the present study aims to validate the effects of orally administered on the perception of time-to-collision of threatening and non-threatening stimuli. To this end, healthy individuals will undergo a double-blind, between-subjects, placebo-controlled pharmaco-eye-tracking experiment and receive a single oral dose of vasopressin (20 IU) or placebo before performing a looming visual stimuli task 45 minutes after administration. The task paradigm will encompass threatening (butterfly, rabbit) and non-threatening (spider, snake) stimuli

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects who volunteer to participate and are able to fully understand and agree with this study by written informed consent.
* Normal or corrected-normal version

Exclusion Criteria:

* History of neuropsychiatric diseases.
* History of cardiac disease, including arrhythmias, aortic stenosis, or congestive heart failure; history of syncope or unexplained loss of consciousness.
* History of hepatic diseases, including cholestasis, biliary obstructive disease, or severe liver dysfunction.
* History of renal diseases, including renal stones or renal failure.
* History of hyponatremia(Serum sodium <135mmol/L) or hyperkalemia (Serum potassium>5.5mmol/L); history of diabetes mellitus or diabetes insipidus
* Known hypersensitivity or allergic reaction to any medication or hormone; strong allergic reaction to food.
* Infections such as COVID-19 or influenza, or unexplained fever.
* Subjects with hypertension (BP ≥130/80mmHg) or hypotension (BP ≤ 90/60mmHg).
* History of alcohol or drug abuse; smoker (≥ 10 cigarettes or ≥ 3 cigars or ≥ 3 pipes/day); smoker using e-cigarettes.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Ratio of judged-time-to-collision to actual-time-to-collision for threatening versus non-threatening stimuli after oral vasopressin administration | 75 minutes - 105 minutes after treatment
  Comparison of the ratio between the judged time to collision and the actual time to collision between the treatment groups for threatening (spider, snake) and non-threatening (rabbit, butterfly) stimuli.

SECONDARY OUTCOMES:
First saccade latency(ms) for threatening versus non-threatening stimuli after oral vasopressin administration | 75 minutes - 105 minutes after treatment
  Comparison of first saccade latencies between treatment groups for threatening (spider, snake) and non-threatening (rabbit, butterfly) stimuli.
Fixation duration(ms) for threatening versus non-threatening stimuli after oral vasopressin administration | 75 minutes - 105 minutes after treatment
  Comparison of mean fixation durations between treatment groups for threatening (spider, snake) and non-threatening (rabbit, butterfly) stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, Dr, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China